CLINICAL TRIAL: NCT03668691
Title: Clinical Outcomes of Joint Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: St. Helena Hospital Coon Joint Replacement Institute (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2016-09-28; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; medial unicompartmental; lateral unicompartmental; bicompartmental; patellofemoral
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Robotic-arm assisted partial knee arthroplasty — Robotic-arm assisted medial unicompartmental knee arthroplasty, lateral unicompartmental knee arthroplasty, bicompartmental knee arthroplasty, patellofemoral knee arthroplasty implants. A robotic arm assisted unicompartmental or bicompartmental knee arthroplasty procedure to replace the medial or lateral and /or patellofemoral compartments of the knee.

SUMMARY:
The purpose of this study is to document the clinical outcomes of partial knee replacement surgery using robotic-arm assisted knee joint surgery at 3 weeks, 6 weeks, 12 weeks, 6 months, 1 year, 2 years, 5 years and 10 years post operative.

DETAILED DESCRIPTION:
The purpose of this study is to document the clinical outcomes of partial knee replacement surgery using robotic-arm assisted knee joint surgery at 3 weeks, 6 weeks, 12 weeks, 6 months, 1 year, 2 years, 5 years and 10 years post operative.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 21 years of age who require a primary robotic-arm assisted unicompartmental knee arthroplasty or bicompartmental knee arthroplasty. These patients will have failed non-operative management of their joint disease and are candidates for partial joint replacement because of pain and stiffness that interferes with their performances or normal daily activities.

Exclusion Criteria:

* Patient had an active infection
* Onlay implants were implanted without bone cement
* Patient does not have enough bone stock to allow for insertion and fixation of the components
* Patient does not have sufficient soft tissue integrity to allow for stability
* Patient has a neurological or muscular deformity that did not allow for control of the knee
* Patient will be excluded from participation in the study if they are cognitively unable to answer study questions
* Pregnant women are excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 21 years of age who require a primary robotic-arm assisted partial knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2011-07; Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
% of patients with Revisions | 10 years after surgery
  To assess the revision rate of this patient population

SECONDARY OUTCOMES:
Patient satisfaction rate | 10 years after surgery
  To assess level of patient satisfaction using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Coon, MD, Principal Investigator — St. Helena Hospital Coon Joint Replacement Institute
Locations (1):
- St. Helena Hospital Coon Joint Replacement Institute, St. Helena, California, United States

IPD SHARING:
Plan to Share IPD: No